CLINICAL TRIAL: NCT03745183
Title: Senna Alata Leaf Decoction as a Treatment for Tinea Imbricata in an Indigenous Tribe in Southern Philippines :a Pilot Study
Brief Title: Senna Alata Leaf Decoction as a Treatment for Tinea Imbricata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philippine Dermatological Society (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDS_PGH_2017_002
Record Dates: First submitted 2017-07-10; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Tinea Imbricata
Keywords: tinea imbricata; Senna alata

STUDY DESIGN:
Intervention Model Description: This study is a preliminary open label, single arm, before and after clinical trial, that utilized Akapulko (Senna alata),a medicinal plant, leaf decoction in the treatment of tinea imbricata. Enrolled, who were recruited during the outreach mission were taught how to make a community-prepared akapulko decoction and were asked to apply it as a leave-on body wash once a day for 28+/-3 days.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Senna alata leaf decoction (Experimental): The participants were instructed to take a bath once a day using a syndet bar and to towel dry their skin before applying the akapulko decoction. Fresh decoction was prepared by the patients every day. After a bath, the patient applied the fresh cooled decoction by hand on the whole body especially on the affected areas and left it to dry. Approximately one glassful (350ml) of akapulko decoction should be consumed for one whole body application. The total duration of daily application should be 4 weeks (28 days +3) until the next outcome assessment.The patients were given illustrated, laminated instructional materials and a tabulated checklist of instructions on how to prepare and apply the decoction which served as a monitoring sheet of each patient.
  Interventions: Other: Senna alata leaf decoction

INTERVENTIONS:
Other: Senna alata leaf decoction — Preparation of the akapulko decoction
  1. Remove the leaflets from the rachis of a mature leaf.
  2. Wash the mature leaflets thoroughly to remove dust, dirt and debris.
  3. In the clay, enamel, or stainless steel pot, place one glassful of closely packed chopped leaves (350 ml glass) and add 2 glasses (around 700ml) of clean water . Use the same glass for measuring the leaves and water.
  4. Cook the leaves and bring to a rolling boil.
  5. When the fluid is reduced to half, remove the decoction from the fire and cool slightly.
  6. Strain the mixture using cheesecloth and press the cut leaves in the strainer to make sure to get as much liquid out of them.
  7. Place the liquid in a clean container (bottle/jar with cover). Label the container clearly as "Akapulko".

SUMMARY:
Background: Tinea imbricata ("tokelau") is a rare form of tinea corporis which is caused by Trichophyton concentricum. It is endemic among the T'boli tribe in Sarangani, Philippines . Temporary remissions, despite antifungal treatment, can be attributed to factors such as genetic susceptibility, widespread poverty, poor hygienic conditions and overcrowding. Limited access to commercial antifungal medications makes the treatment of tinea imbricata a pressing public health concern.

Senna alata grows abundantly in the areas where the T'boli tribe resides. Anecdotal reports about its efficacy as a treatment for tinea imbricata exist and need to be further validated.

Objective: This study aims to assess the efficacy and safety of a community-prepared Senna alata leaf decoction in the treatment of tinea imbricata.

Methods: This study is a preliminary open label, before and after clinical trial. Enrolled patients were taught how to make Senna alata leaf decoction and were asked to apply it as a leave-on body wash once a day for 28+/-3 days. Disease severity, pruritus visual analogue scale scores (VAS) and potassium hydroxide smear (KOH) of the skin scrapings were evaluated before and after treatment. Two separate assessors evaluated post treatment severity based on standard photographs. Diagnostic concordance was determined using Cohen's kappa statistics. Wilcoxon paired signed-rank test was used to analyzed before and after clinical parameter scores. Adverse drug events were recorded.

DETAILED DESCRIPTION:
Introduction:

Tinea imbricata is a rare form of tinea corporis caused by Trichophyton concentricum, an anthropophilic dermatophyte. Its lesions would present embossed "maze-like" or lace-like pattern of embosed concentric rings mainly on the trunk and extensor surfaces of both extremities, sparing the palms, soles, hair and nails. Due to the rarity of the disease, limited epidemiologic and prevalence studies exist. (Halickova, 2008) Tine imbricata is known to be endemic in places such as the Paciﬁc Islands of Oceana, South East Asia, India, Sri-Lanka, North, Central and South America. (Halickova, 2008 and Pihet, 2008) The first case was discovered in the southern Philippines by William Dampier in 1789. (Fernandez, 1962) In 2010, cases of tinea imbricata were found to still exist among T'boli tribe who live in the mountainous areas of Kiamba in Sarangani through the University of the Philippines- Department of Science and Technology (UP-DOST) telemedicine project. (Carpio, 2010) The inherited susceptibility of T.concentricum infection may explain why the disease affects only specific group of people. The most accepted inheritance pattern is autosomal recessive attributing to the inherited defect in cell-mediated immunity, which results to failure of the T-lymphocytes to become sensitized to the fungi and mount an immune response. Majority of the patients are blood-related individuals and rarely infect unrelated individuals even after close contact or cohabitation., Other risk factors are isolated and primitive living conditions especially in humid areas, widespread poverty, poor hygienic conditions and overcrowding. (Bonifaz, 2003 and Bonifaz, 2004) Antifungals are the mainstay treatment against Trichophyton concentricum. Griseofulvin, 500 mg/tab twice daily, and terbinafine, 250 mg once daily, for at least 4 weeks result to complete resolution. (Wingfield, 2004) However, these commercial antifungal preparations are costly and not readily available in the health centers of Sarangani. Furthermore, even with systemic antifungal intake, disease remission would only last for at least 8 weeks post-treatment. Alternative treatment options that will promote clearance of the infection that are accessible, inexpensive and practical to use should be explored.

Antifungals from local plant sources are one of the potential alternatives. Among these, Senna alata has validated efficacy on superficial dermatophytic infections and is included in the Philippine National Drug Formulary. It is a tropical ornamental shrub, also known as candle bush and locally as "Akapulko, which grows throughout the low and medium altitude areas of the country including Sarangani.

Chemical screening of the leaves and roots of S. alata revealed the anthraquinones and its derivatives such as aloe, emodin, chrysophanol, and rhein, are the major components responsible for its antifungal activity. These are naturally occurring phenolic compounds are readily oxidized to form a phenolate ion or quinone, which aids in the scavenging and entrapment of microorganisms. Furthermore, phenols impair a variety of enzyme systems that are involved in the microorganism's energy production. They also disrupt the integrity of the cell membrane and interfere with the synthesis of its structural components. (Hemen and Ledwani,2012) There were anecdotal reports on the efficacy of akapulko decoction against tinea imbricata. A decoction is the liquid resulting from concentrating the essence of the substance by heating or boiling, especially a medicinal preparation made from a plant. Plant parts such as leaves can be used in decoctions. The first anecdotal report was published by Dofitas and Non last 2010. Senna alata leaf decoction was used as leave-on body wash in a T'boli woman resulting in complete clearance of the lesions. In the case series by Carpio et. al., S. alata leaf decoction resulted to partial improvement of the skin lesions. (Dofitas and Non, 2010 and Caprio, 2010) At present there are no existing clinical trials about the use of akapulko as an alternative or complementary treatment to tinea imbricata. The favorable results from the anecdotal and case series studies pave the way for the consideration of akapulko decoction as a part of an accessible and affordable treatment regimen for tinea imbricata.

II Objectives:

General objectives: This study aims to assess the efficacy and safety of Senna alata leaf decoction applied once daily in the treatment of tinea imbricata.

Specific objectives:

1. To determine the treatment response at the end of four weeks (28 days +/-3) as measured by disease severity, pruritus visual analogue scale score and potassium hydroxide smear conversion of the patients with tinea imbricata treated once daily with Senna alata leaf decoction
2. To document the adverse reactions associated with Senna alata leaf decoction application.

III Methods:

This study was a preliminary open label, before-and after clinical trial. This study took place at Kiamba Municipality, Sarangani Province, Mindanao from November 2014 to January 2015. The duration of patient involvement was 4 weeks (28+3 days). Figure 1 shows the flow chart of the study procedure.

Recruitment of participants: An outreach skin clinic, manned by dermatology residents and consultants of the University of the Philippines- Philippine General Hospital, was conducted in the local health center. Patients with any skin disease and suspected tinea imbricata cases were invited to consult. Patient recruitment began during the outreach mission and was continued even thereafter. A consultant investigator assessed eligibility and disease severity of the participants, during and even after the outreach mission. Trained research assistants collected skin scrapings from active skin lesions of patients.

Each participant was assigned code numbers written on the case record forms. The participants' names with the corresponding numbers were recorded in a separate registry.

Securing consent and enrolment of participants: All patients with clinically diagnosed tinea imbricata and with microscopically positive KOH smear were invited by the investigators to join the study. The purpose, duration, benefits and possible adverse effects were explained to all participants and signed consent forms were secured by research assistants who could speak T'boli dialect. A thumb mark was obtained in place of a signature for illiterate participants. (Appendices A, B, and C)

Enrolled patients were subjected to the following steps before starting therapy:

1. Detailed history-taking and physical examination
2. Collection of skin scrapings and microscopic confirmation of fungal elements in skin scrapings using potassium hydroxide mount
3. Accomplishment of the standard case record forms, which details the severity of the disease, pruritus VAS score and adverse drug effects. (Appendix D)
4. Pre-treatment photographic documentation. A written consent was obtained prior to photographic documentation of each patient. Photography was done in a private room.

Application of Akapulko leaf decoction:

The participants were instructed to take a bath once a day using a syndet bar and to towel dry their skin before applying the akapulko decoction. Fresh decoction was prepared by the patients every day. After a bath, the patient applied the fresh cooled decoction by hand on the whole body especially on the affected areas and left it to dry. Approximately one glassful (350ml) of akapulko decoction should be consumed for one whole body application. The total duration of daily application should be 4 weeks (28 days +3) until the next outcome assessment.

The patients were given illustrated, laminated instructional materials and a tabulated checklist of instructions on how to prepare and apply the akapulko decoction. This served as a monitoring sheet of each patient. (Appendix E) The barangay health workers underwent hands-on training by the investigators on the preparation of the akapulko leaf decoction. Trained research assistants conducted demonstration of the akapulko preparation to the enrolled patients. (Appendix F)

Clinical Parameters: Each patient was assessed based on disease severity based on erythema, scaling and area of involvement. (Tables 1-3) Then, composite scores were combined and graded no disease, mild, moderate and severe. (Table 4) Pruritus severity was gauge using 10-cm pruritus visual analogue scale score. KOH smear of skin scrapings was also done before and after treatment.

Outcome assessment:

Clinical response to treatment was assessed after 4 weeks. Standard photographs were taken by the research assistants for documentation and sent electronically via email to the investigators. A panel of two dermatologists who had prior clinical experience with tinea imbricata assessed the treatment response based on the digital photographs taken at the end of the treatment period. Post-treatment VAS scores were recorded.

Mycologic cure was assessed as a negative KOH mount after 1 month of treatment in both treatment groups. The research aides or the public health nurse collected skin scrapings for KOH on the same site as the pre-treatment KOH source. Samples were placed in clean pieces of folded bond paper inside a properly sealed envelope and airmailed to the investigators for KOH microscopic examination.

Data management and analysis A standard case record form was used to collect patient data (Appendix A). Accomplished records were checked for accuracy and completeness by the investigators in the field. Data gathered were encoded in an electronic spreadsheet, Microsoft Excel 2011.

Descriptive analysis was done, which included epidemiologic characteristics, initial disease severity, and clinical outcome per patient. Clearance rates were computed after 4 weeks using the formulas below.

Clearance rate = Number of patients who underwent clearance x 100/ Total number of patients enrolled

Partial clearance rate = Number of patients who underwent partial clearance X 100/Total number of patients enrolled

Failure rate = Number of patients who had no improvement + worsening disease severity X100/Total number of patients enrolled

Each patient was classified as with complete clearance, partial clearance or no clearance. Subgroup analysis by disease severity was performed. Diagnostic concordance between the two consultants who assessed disease severity was determined using Cohen's kappa statistics. Wilcoxon paired signed rank test was used to analyzed before and after clinical parameter scores. Adverse drug events, reported by the patients, were recorded as a frequency distribution.

Adverse reactions Presence of any adverse reactions was noted. Subjects were instructed to report side effects for proper management. (Table 5) Participants with mild to severe adverse drug effects were to be withdrawn from the study and provided appropriate management by the investigators.

Ethical considerations:

This study was conducted in accordance to the guidelines of the Helsinki declaration. The study protocol was formulated in accordance to the guidelines imposed by the National Ethical Guideline for Health Research published by the Philippine Health Research Ethics Board and was conducted upon the approval of the institution's ethics review board. Since indigenous people are involved as subjects, this study was approved the National Commission on Indigenous People (NCIP). A research grant was received from the Philippine Dermatological Society. There were no conflicts of interest in the conduct of this research.

ELIGIBILITY:
Inclusion Criteria:

1. Indigenous T'boli patient aged 18 years old and above, male or female
2. Patients with clinically diagnosed tinea imbricata with microscopically confirmed skin scraping positive for potassium hydroxide (KOH)

Exclusion Criteria:

1. Patients who were treated or undergoing treatment with topical anti-fungal for 2 weeks or oral anti-fungal 1 month before the study
2. Patients who were taking other systemic medications such as cytotoxic and immunosuppressive drugs
3. Patients with known liver disease, kidney dysfunction, hematologic problems (e.g. anemia)
4. Patients with or suspected allergy to Senna alata extract

The participation of the subjects were completely voluntary. Participants were allowed to withdraw from the study at anytime and for any reason without prejudice to their subsequent medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
Improvement in disease severity | Before and after the treatment period of 1 month
  Disease severity was measured by body surface area of involvement, erythema and scaling . After which, their composite scores were combined and graded no disease, mild, moderate and severe.
  Body surface area of involvement grading Score Characteristic 0 No lesions
  1. Lesions occupy an aggregate surface area less than or equal to 5cm x 5cm
  2. Aggregate surface area greater than 5cm x 5cm but less than 10cm x 10cm
  3. Aggregate surface area of greater than 10cm x 10cm
  Erythema grading Score Characteristic 0 No erythema
  1. Nearly imperceptible erythema
  2. Moderate erythema (pinkish skin)
  3. Intense erythema
  Scaling grade Score Characteristic 0 No scaling
  1. Fine white scales
  2. Moderate scales
  3. Large scales
  Composite Scores Category Score No disease 0 Mild For composite score of 1-3 Moderate For composite score of 4 -6 Severe For composite score of 7- 9

SECONDARY OUTCOMES:
Adverse Events | Before and after the treatment period of 1 month
  Presence of adverse drug effects were noted. Subjects were instructed to report to the research assistants or to the local health center in case any of these adverse drug events occurred for proper management. Participants with mild to severe adverse drug effects were withdrawn from the study and provided appropriate management by the investigators.

OTHER OUTCOMES:
Improvement in pruritus visual analogue scale scores | Before and after the treatment period of 1 month
  The visual analogue scale is a 10-cm long line oriented horizontally or vertically used to indicate the patient's intensity of pruritus by crossing the line at the point the corresponds to the patient's pruritus severity. The patients' pruritus was assessed using the VAS scale in which the patients were instructed to select a point along the 10-cm line for his/her assessment, with "0" meaning no pruritus and "10" meaning the most severe pruritus they can imagine.
potassium hydroxide smear conversion | Before and after the treatment period of 1 month
  Potassium hydroxide mount (KOH) test of the lesions were done before , where in KOH 10% reagent dropped on the skin scales to confirm the presence of fungal infection by microscopic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E Alpapara, MD, Principal Investigator — Philippine Dermatological Society; Belen L Dofitas, MD, Study Director — Philippine Dermatological Society

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pihet M, Bourgeois H, Maziere JY, Berlioz-Arthaud A, Bouchara JP, Chabasse D. Isolation of Trichophyton concentricum from chronic cutaneous lesions in patients from the Solomon Islands. Trans R Soc Trop Med Hyg. 2008 Apr;102(4):389-93. doi: 10.1016/j.trstmh.2008.01.002. Epub 2008 Mar 4. PMID 18295290
- [Background] FERNANDEZ MC, JAO RL. Tinea imbricata successfully treated with griseofulvin. Report of a case. Arch Dermatol. 1962 Jul;86:65-7. doi: 10.1001/archderm.1962.01590070071011. No abstract available. PMID 13892414
- [Background] Havlickova B, Czaika VA, Friedrich M. Epidemiological trends in skin mycoses worldwide. Mycoses. 2008 Sep;51 Suppl 4:2-15. doi: 10.1111/j.1439-0507.2008.01606.x. PMID 18783559
- [Background] CHERMSIRIVATHANA S, BOONSRI P. A case of tinea imbricata (Hanumarn ringworm) treated with fulcin. Aust J Dermatol. 1961 Jun;6:63-6. doi: 10.1111/j.1440-0960.1961.tb01331.x. No abstract available. PMID 13878721
- [Background] Bonifaz A, Araiza J, Koffman-Alfaro S, Paredes-Solis V, Cuevas-Covarrubias S, Rivera MR. Tinea imbricata: autosomal dominant pattern of susceptibility in a polygamous indigenous family of the Nahuatl zone in Mexico. Mycoses. 2004 Aug;47(7):288-91. doi: 10.1111/j.1439-0507.2004.00989.x. PMID 15310331
- [Background] Bonifaz A, Archer-Dubon C, Saul A. Tinea imbricata or Tokelau. Int J Dermatol. 2004 Jul;43(7):506-10. doi: 10.1111/j.1365-4632.2004.02171.x. PMID 15230889
- [Background] Hemen, Dave and Ledwani, Lalita. A review on anthraquinones isolated from Cassia species and their applications. Indian Journal of Natural Products and Resources. September 2012. Vol. 3 (3), pp.291-319
- [Background] Núñez Montoya, S.C., Comini L.R., and Cabrera J.L.. Antimicrobial activity of natural photosensitizing anthraquinones. Science against microbial pathogens: communicating current research and technological advances. Department of Pharmacology. 2011. pp 3-13
- [Background] Okwu, D.E. and Nnamdi, F.U.Cannabinoid Dronabinol alkaloid with antimicrobial activity from Cassia alata Linn. Der Chemica Sinica. 2011. Vol 2(2): 247-254
- [Background] Philippine Health Research Board. National Ethical Guidelines for Health Research. 2011.pp 54-58 and 91-96.
- [Background] National Administrative Order No. 3 " The Revised Guidelines and Prior Informed Consent (FPIC) and Related Processes f 2012"
- [Background] Duke, James. Duke's Handbook of Medicinal Plants of the Bible. USA: CRC Press, 2007.
- [Result] Wingfield AB, Fernandez-Obregon AC, Wignall FS, Greer DL. Treatment of tinea imbricata: a randomized clinical trial using griseofulvin, terbinafine, itraconazole and fluconazole. Br J Dermatol. 2004 Jan;150(1):119-26. doi: 10.1111/j.1365-2133.2004.05643.x. PMID 14746625
- [Result] Dofitas BL and Non BL., Tinea Imbricata: Case Series on Three Patients in Sarangani, Philippines. Acta Medica Philippina. 44(3). (2010)
- [Result] Carpio, V , Dofitas, B and Frez, L. (2010). Blekis: Tinea imbricata in Sarangani, Philippines.Unpublished manuscript.
- Available data/document: Study Protocol — https://drive.google.com/open?id=1ial1puH4ar075LyGcoWIrU1AXclt3FO-
- Available data/document: Tables 1-5 — https://drive.google.com/open?id=1pmZyUhTfoOPWRDJgEFjMsa_K9bvQ_Lon
- Available data/document: Figure 1. Flow chart of the study procedure — https://drive.google.com/open?id=1MpUGMeNkzeOlThYZ_Zur4xTgt5cOvQNN
- Available data/document: Informed Consent Form — https://drive.google.com/open?id=1kV91jvmtUDi_BA2paf-iszXb7bCnKHZO
- Available data/document: Individual Participant Data Set — https://drive.google.com/open?id=1n3y-FDFc63KGyGfbkNBlpLJ-6HE9BBUZ
- Available data/document: Appendix E. Illustrated checklist for the T'boli — https://drive.google.com/open?id=1t2b-wyQsJaTEy6qqJCiL4Opg-Hdvdxzj
- Available data/document: Appendix F. Illustrated instruction on Senna alata decoction preparation — https://drive.google.com/open?id=17hMRr2-GhROnq7Gdw0Skd1KFApCpCgzy